CLINICAL TRIAL: NCT04375384
Title: Pilot Phase II Study to Evaluate Effect of Cetuximab Given as Single Agent After Immunotherapy With PD-1 Inhibitors in Patients With Head and Neck Squamous Cell Carcinoma
Brief Title: Cetuximab After Immunotherapy for the Treatment of Head and Neck Squamous Cell Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00065239; WFBCCC 60220 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Metastatic Head-and-neck Squamous-cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cetuximab (Experimental): Patients receive cetuximab IV over 60-120 minutes once every week in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cetuximab; Other: Questionnaire administration; Other: Quality of life assessment

INTERVENTIONS:
Drug: Cetuximab — A loading dose of Cetuximab will be administered intravenously in the first day of treatment. The dose is 400 mg/m2 and will be infused over 2h followed by 1h observation.
  The maintenance dose of Cetuximab is 250 mg/m2 and will be infused over 1h. No further observation time needed.
  The maintenance dose of cetuximab will be given every 7 days (+/- 2 days) starting 7 days (+/- 2 days) after the loading dose of cetuximab.
  Pre-medicate with 50 mg Diphenhydramine IV before the loading dose of Cetuximab and as per standard of care before the maintenance treatment.
Other: Questionnaire administration — Ancillary studies
Other: Quality of life assessment — Ancillary studies

SUMMARY:
This is a Phase II treatment, non-randomized, open label clinical trial to study the efficacy of the Cetuximab when administered as single agent in recurrent/ metastatic head and neck squamous cell carcinoma after the failure or intolerance of immuno-oncology or immuno-oncology combined with chemotherapy.

DETAILED DESCRIPTION:
Primary Objective:

• To measure Overall Response Rate to treatment with Cetuximab as single agent in patients with recurrent or metastatic head and neck squamous cell cancer who failed PD-1 inhibitors alone or in combination with chemotherapy.

Secondary Objective(s):

* Measure Duration of Response (DUR), Progression Free Survival and Overall Survival and for treatment with single agent Cetuximab after immunotherapy with PD-1 inhibitors in Head and Neck Squamous Cell Carcinoma.
* Evaluate treatment toxicity with single agent Cetuximab in this patient population.

OUTLINE: Patients receive cetuximab intravenously (IV) over 60-120 minutes once every week in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 week and then every 6-8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed head and neck squamous cell carcinoma.
* Measurable disease by scans- at least one measurable lesion.
* Patients must have received previous treatment with immunotherapy with PD-1 inhibitor alone or in combination with chemotherapy.
* Patients must have a Performance Status of 0-2.
* Patients must be greater than or equal to 18 years old.
* Participant is willing and able to comply with the protocol for the duration of the study.
* Ability to understand and the willingness to sign an Institutional Review Board-approved informed consent document.

Exclusion Criteria:

* Prior treatment with Cetuximab or prior therapy that specifically and directly targets the epidermal growth factor receptor (EGFR) pathway in the last five (5) days.
* Prior allergic reaction to Cetuximab.
* History of allergic reactions attributed to compounds of chemical or biologic composition similar to those of Cetuximab.
* Patients receiving any other investigational agents.
* Patient is on medications that need to be continued and that might interact with Cetuximab.
* Any uncontrolled condition, which in the opinion of the investigator, would interfere in the safe and timely completion of study treatment and procedures.
* Participant with a history of interstitial lung disease (e.g. pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on screening chest imaging.

Any of the following conditions:

* Serious or non-healing wound, ulcer, or bone fracture at the discretion of treating physician
* history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of study enrollment
* history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study enrollment
* history of myocardial infarction, ventricular arrhythmia, stable/unstable angina, -symptomatic congestive heart failure, coronary/peripheral artery bypass graft or stenting or other significant cardiac disease within 6 months prior to study enrollment
* history of arterial or venous thrombosis/thromboembolic event, including pulmonary embolism within 6 months of study enrollment
* any condition requiring the use of immunosuppression, excluding rheumatologic conditions treated with stable doses of corticosteroids.

Pregnancy, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Overall Response Rate To Treatment with Cetuximab | 14 days before start of treatment, 7 weeks after start of treatment, and then every 6-8 weeks for the duration of treatment, up to approximately 2 years.
  Overall response rate is defined as the proportion patients achieving partial response or complete response per RECIST v1.1 criteria. An estimate of a 95% Exact Clopper Pearson confidence interval will be used. RECIST 1.1 criteria will be used to measure tumor size: Measurable disease is defined by the presence of at least 1 measurable lesion. A lesion, not previously irradiated per the protocol prior to enrollment, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with CT or MRI and that is suitable for accurate repeated measurements. Non-measurable: All other lesions, including small lesions (longest diameter <10 mm or pathological lymph nodes with ≥10 mm to <15 mm short axis at baseline). Only participants with measurable disease at baseline will be included in the study.

SECONDARY OUTCOMES:
Duration of Progression Free Survival | At 6 months and at 1 year after enrollment on study
  Progression free survival will be defined as progression of local-regional disease, distant metastases or death without progression and will be reported as median progression-free survival as well as progression free survival at 6 month and 1 year time points. Investigators will estimate Kaplan Meier survival curves and estimate the median duration of response with 95% confidence intervals for these measures.
Duration of Overall Survival | At 6 months and at 1 year after enrollment on study
  Overall survival is defined as death due to any cause and will be reported as median overall survival as well as overall survival at 6 month and 1 year time points. Investigators will estimate Kaplan Meier survival curves and estimate the median duration of response with 95% confidence intervals for these measures.
Duration of Response | At 6 months and at 1 year after enrollment on study
  Response is defined as (failure - progression of loco-regional disease or distant metastasis) Investigators will estimate Kaplan Meier survival curves and estimate the median duration of response and will also estimate 95% confidence intervals for this measure.
Number of Treatment-Related Toxicities with Cetuximab as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 2 years
  Treatment-related side effects will be collected before each treatment based on clinical laboratory and radiologic changes and will be graded and reported. All patients who receive at least one dose of cetuximab will be considered evaluable for safety analysis. Investigators will create frequency tables that count the number and severity of toxicities observed in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Porosnicu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burcher KM, Bloomer CH, Gavrila E, Kalada JM, Chang MJ, Gebeyehu RR, Song AH, Khoury LM, Lycan TW, Kinney R, D'Agostino R Jr, Bunch PM, Shukla K, Triozzi P, Furdui CM, Zhang W, Porosnicu M. Study protocol: phase II study to evaluate the effect of cetuximab monotherapy after immunotherapy with PD-1 inhibitors in patients with head and neck squamous cell cancer. Ther Adv Med Oncol. 2024 Jan 19;16:17588359231217959. doi: 10.1177/17588359231217959. eCollection 2024. PMID 38249330